CLINICAL TRIAL: NCT00789295
Title: Mediterranean vs. Low-Carbohydrate Diet : Which is the Best Dietary Approach for Treating Postprandial Lipid Abnormalities and Improving Glucose Control in Type 2 Diabetic Patients?
Brief Title: Mediterranean Diet and Postprandial Lipemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Angela A. Rivellese, MD, Department of Clinical and Experimental Medicine Federico II University Naples
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 29102008
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2008-11-11 (Estimated); Status verified 2008-10

CONDITIONS: Postprandial Lipemia; Type 2 Diabetes
Keywords: Mediterranean diet; Postprandial lipids; Postprandial glucose; High fibre diet; Low- CHO diet; High MUFA diet; Dietary approach
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mediterranean diet (Active Comparator): The Mediterranean diet: relatively rich in Carbohydrate(52% of the total daily energy intake), rich in dietary fibre (28g/1000 kcal both of soluble and unsoluble types) and with a low glycemic index (51%)
  Interventions: Other: Mediterranean diet and Low-Carbohydrates diet
- Low-Carbohydrates diet (Active Comparator): Low-carbohydrates diet : diet rich in MUFA (23%), relatively low in CHO (45%), low in dietary fibre (8g/1000 kcal) and with a relatively high glycemic index (87%)
  Interventions: Other: Mediterranean diet and Low-Carbohydrates diet

INTERVENTIONS:
Other: Mediterranean diet and Low-Carbohydrates diet — The Mediterranean diet: relatively rich in Carbohydrate(52% of the total daily energy intake), rich in dietary fibre (28g/1000 kcal both of soluble and unsoluble types) and with a low glycemic index (51%) versus Low-carbohydrates diet : diet rich in MUFA (23%), relatively low in CHO (45%), low in dietary fibre (8g/1000 kcal) and with a relatively high glycemic index (87%)for 4 weeks

SUMMARY:
The aim of this intervention study was to evaluate in type 2 diabetic patients the effects on postprandial lipemia and other metabolic parameters (in both everyday life conditions and after a standard test meal) of two diets, one moderately rich in CHO, rich in fibre and with a low glycemic index (Mediterranean diet), and the other low in CHO and rich in MUFA (Low-CHO diet).Since adipose tissue, mainly through its lipolytic activities, is considered as having a pivotal role in the regulation of postprandial lipid metabolism, a further aim of our study was to clarify the role of adipose tissue in modulating the postprandial lipid response induced by the two dietary approaches by evaluating the activities of lipoprotein lipase (LPL) and hormone-sensitive lipase (HSL).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Stable metabolic control (HbA1c<8.0%) on diet or diet alone or diet+metformin
* BMI<30 kg/m2 and body weight stable during the last six months.
* Both sexes; only post-menopausal women.
* Normal fasting lipid levels
* No use of hypolipidemic drugs

Exclusion Criteria:

* Patient with renal (serum creatinine >1.5 mg/dl) or hepatic (serum transaminases >three times upper normal values) impairment.
* Patients with history of cardiovascular disease.
* Pre-menopausal women.
* Any other acute or chronic degenerative disease.
* Anemia (Hb<12 g/dl).
* Uncontrolled blood pressure.
* Use of any drugs able to interfere with the study medications

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-03

PRIMARY OUTCOMES:
Postprandial response triglyceride of chylomicrons and large VLDL | 4 weeks

SECONDARY OUTCOMES:
Blood glucose and insulin response to test meal | 4 weeks
Lipolytic activities | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Riccardi, Prof, Study Chair — Department of Clinical and Experimental Medicine, Federico II University Hospital, Naples, Italy
Locations (1):
- Department of Clinical and Experimental Medicine, Federico II University Hospital,, Naples, Naples, Italy

REFERENCES:
- [Background] Rivellese AA, De Natale C, Di Marino L, Patti L, Iovine C, Coppola S, Del Prato S, Riccardi G, Annuzzi G. Exogenous and endogenous postprandial lipid abnormalities in type 2 diabetic patients with optimal blood glucose control and optimal fasting triglyceride levels. J Clin Endocrinol Metab. 2004 May;89(5):2153-9. doi: 10.1210/jc.2003-031764. PMID 15126535
- [Background] Lopez-Miranda J, Williams C, Lairon D. Dietary, physiological, genetic and pathological influences on postprandial lipid metabolism. Br J Nutr. 2007 Sep;98(3):458-73. doi: 10.1017/S000711450774268X. PMID 17705891
- [Background] Lairon D, Play B, Jourdheuil-Rahmani D. Digestible and indigestible carbohydrates: interactions with postprandial lipid metabolism. J Nutr Biochem. 2007 Apr;18(4):217-27. doi: 10.1016/j.jnutbio.2006.08.001. Epub 2006 Oct 31. PMID 17079126
- [Derived] De Natale C, Annuzzi G, Bozzetto L, Mazzarella R, Costabile G, Ciano O, Riccardi G, Rivellese AA. Effects of a plant-based high-carbohydrate/high-fiber diet versus high-monounsaturated fat/low-carbohydrate diet on postprandial lipids in type 2 diabetic patients. Diabetes Care. 2009 Dec;32(12):2168-73. doi: 10.2337/dc09-0266. Epub 2009 Sep 9. PMID 19741188